CLINICAL TRIAL: NCT04357912
Title: Utilizing Activity Trackers to Promote Physical Activity in People With Epilepsy: Can we Make a Difference?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Neurological Society Research Grant-2020 (Unknown)
Responsible Party: Principal Investigator, Katherine Marie Johns Harris, Clinical Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-20-0173
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Epilepsy
Keywords: epilepsy; exercise; activity tracker
MeSH Terms: conditions — Epilepsy; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Behavioral: Activity Tracker Group
- Control Group (Active Comparator)
  Interventions: Behavioral: Standard of Care Group

INTERVENTIONS:
Behavioral: Activity Tracker Group — In addition to the standard of care exercise education, participants in the activity tracker group will be provided a Fitbit physical activity tracker at no cost to the participants. They will be asked to download the Fitbit application (app) to their personal smartphone device to allow them to see their own data collected by the Fitbit. They will also be asked to download the Stridekick app for the purpose of sharing their activity tracker data electronically with the study team and having the opportunity to participate in fitness challenges through the app. App accounts will be created by the participants with usernames that do not contain the participant's identifiable personal information. Optional fitness challenges will be created once per month by the study investigators, and participants will also receive a weekly message of encouragement from the study team.
  Arms: Experimental group
Behavioral: Standard of Care Group — Participants will receive standard of care exercise education.
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate standard of care exercise education alone or in combination with a wearable physical activity tracker in people with epilepsy (PWE) to determine the most effective way to increase physical activity and measure impact on depression, anxiety, quality of life, sleep, and seizure frequency.

ELIGIBILITY:
Inclusion Criteria:

* patient of the Texas Comprehensive Epilepsy Program at UTHealth-McGovern Medical School
* diagnosis of epilepsy
* be able to provide consent in English
* complete surveys independently
* be able to sync Fitbit data

Exclusion Criteria:

* currently using a wearable physical activity tracker prior to enrollment
* pregnant or planning to become pregnant during the study duration
* planning to undergo epilepsy surgery during the study duration

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Number of steps taken by participant | 3 months after enrollment
Total distance traveled by participant | 3 months after enrollment
Total time participant is active | 3 months after enrollment
  measured in minutes

SECONDARY OUTCOMES:
Depression as measured by the Patient Health Questionnaire depression scale (PHQ-9) | Baseline
  this is scored form 0-27 with a higher number indicating higher severity
Depression as measured by the Patient Health Questionnaire depression scale (PHQ-9) | end of study (3 months after enrollment)
  this is scored form 0-27 with a higher number indicating higher severity
Anxiety as measured by the General Anxiety Disorder 7-item scale (GAD-7) | Baseline
  The GAD-7 score ranges form 0 (minimal anxiety) to 21 (severe anxiety)
Anxiety as measured by the General Anxiety Disorder 7-item scale (GAD-7) | end of study (3 months after enrollment)
  The GAD-7 score ranges form 0 (minimal anxiety) to 21 (severe anxiety)
Sleep as measures by the Epworth Sleepiness Scale (ESS) | Baseline
  The ESS scale ranges form 0 (would never dose) to 3 (high chance of dozing)
Sleep as measures by the Epworth Sleepiness Scale (ESS) | end of study (3 months after enrollment)
  The ESS scale ranges form 0 (would never dose) to 3 (high chance of dozing)
Quality of life as assessed by the Quality of Life in Epilepsy (QOLIE-10-P) survey | Baseline
  The range of total scores for the QOLIE-10-P survey is 1 to 5, with 1 indicating a better outcome.
Quality of life as assessed by the Quality of Life in Epilepsy (QOLIE-10-P) survey | end of study (3 months after enrollment)
  The range of total scores for the QOLIE-10-P survey is 1 to 5, with 1 indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Harris, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No